CLINICAL TRIAL: NCT02583204
Title: Taxane Chemotherapy and Nail Toxicity in Women With Breast Cancer; Stage Two: Evaluation of Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN15ON391
Record Dates: First submitted 2015-09-22; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer; Nail Toxicity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control - standard care (No Intervention): Participants will receive standard care regarding nail toxicity. This entails advice to keep nails trim and the provision of a nail oil to massage into the nail daily. Participants will also receive advice in relation to general healthy living.
- Intervention - Oncolife drops (Experimental): Participants will receive the same standard care as the control arm, except for the nail drops. The participants will also receive Onicolife nail drops to be applied twice daily.
  Interventions: Device: Onicolife nail drops
- Intervention - Nail polish (Experimental): Participants will receive the same standard care as the control arm, except for the nail drops. The participants will also receive a dark coloured nail polish to be applied as instructed.
  Interventions: Other: Nail polish

INTERVENTIONS:
Device: Onicolife nail drops — The prescription free, CE (Conformité Européenne) marked product is for local application, and has a novel mode of action involving the modulation of mast cell action with the fatty acid amide, Adelmidrol ®. Mast cells are known to have a key role in the ability of the body to promote healing /repair and control tissue damage caused by chemo and radiotherapy. This includes damage to the nail and/ or nail matrix. OnicoLife ® thus helps to control inflammation and pain whilst antimicrobial action also provides antibacterial and antifungal support.
  Arms: Intervention - Oncolife drops
Other: Nail polish — One dark colour of nail polish (deep burgundy/red) will be used in this study since this colour is considered more acceptable to many more women than a pure black coloured nail polish and hence, more likely to ensure compliance. No nail polish containing hardeners will be used since there is some evidence to suggest they can induce nail changes. As dark nail polish can stain the nail plate (and therefore mask any changes in nail pigmentation induced by chemotherapy), one clear base coat, two coats of coloured, and one clear top coat of polish will be required for each application. This standard of application is proposed as a gold standard for the prevention of nail staining and hypersensitivity reactions by an eminent podiatrist (Spalding, 2008).
  Arms: Intervention - Nail polish

SUMMARY:
The study compares three strategies to prevent/minimise nail problems occuring in women, with breast cancer, undergoing Taxane chemotherapy. The strategies are: application of nail polish and normal care; application of Onicolife drops and normal care and; normal care only.

DETAILED DESCRIPTION:
This protocol outlines a proposal to investigate whether the use of a dark-coloured nail polish or OnicoLife nail drops, compared to standard care, from commencement of taxane based chemotherapy until three months after completion, is effective in preventing or minimising chemotherapy-induced nail problems.

In the UK, taxane based chemotherapy is used within neo-adjuvant, adjuvant and metastatic settings. Taxotere (docetaxel) is provided in an neo-adjuvant and adjuvant setting every three weeks, taxol (paclitaxel) and taxotere are provided in the metastatic setting either weekly or three weekly.

Taxane based chemotherapy with Taxotere has been shown to improve progression-free, disease free and overall survival in the metastatic setting. TACT, a large phase III adjuvant, open-label randomised controlled trial of sequential taxotere following anthracycline chemotherapy did not show any overall gain from the addition of Docetaxel to standard anthracycline chemotherapy. There are many common side effects associated with chemotherapy such as nausea and vomiting, alopecia and neutropenia but with correct management, these are generally tolerated. There is evidence that while taxane chemotherapy improves clinical response and reduces troublesome side effects such as nausea and vomiting, it is also demonstrated to result in more nail toxicity/ changes than AC (adriamycin-cyclophosamide) therapy (92% versus 32% respectively).

It has been suggested that nail problems associated with chemotherapy are under reported in terms of the incidence and severity. Evidence of chemotherapy-induced nail changes was found in studies that involved randomisation to taxane or non-taxane-containing regimens and /or combination therapy.

Case study reports in oncology journals also highlighted nail toxicity and abnormalities following treatment with taxane therapy and associated challenges with continuation of therapy in breast cancer and patients with lung cancer.

Nail toxicity can occur on some or all of the hands and/ or feet, and may vary in appearance, severity and function. Reported problems vary from pigmentation, discolouration, and thinning or ridging of nails to Beau's lines, Mee's lines, oncycholysis, sub-ungual hyperkeratosis, acute paronchyia, sub-ungual haemorrhage, and loss of nail plate. These are thought caused by the direct effect on the nails from the drugs and is hypothesised as an effect mediated by the drug stabilising chemicals. There is evidence that taxanes appear to stimulate the matrix melanocytes, which the authors suggest as independent of ACTH (adrenocorticotropic hormone), MSH4 (MutS protein homolog 4), and UV (ultraviolet) light. Others suggest taxane-induced thrombocytopenia and vascular abnormalities as a precursor to sub-ungual haematomas and haemorrhagic onycholysis.

Nail changes may appear in temporal relationship with drug intake and vary depending on the structure of the nail affected. Nail toxicities related to chemotherapy are significantly higher in weekly compared to 3-weekly regimens. In one study, more frequent and severe toxic effects occurred in dose-dense regimens than in the standard TEC5 regimen, with grade 3-4 nail changes occurring in 73% of patients receiving EC-T6 therapy. Fifty-eight percent of cancer patients treated with EGFRI developed nail abnormalities, typically after 6-8 weeks of treatment, including paronychia. Cumulative dose in chemotherapy appears significant in the incidence of nail toxicity, the median cumulative dose of the anthracycline doxorubicin, reported as 22.5 mg/m² and mean cumulative dose of taxane docetaxel as 810 mg/m². Most cutaneous/ nail changes have a tendency to develop after a number of treatment cycles, typically after cycle 4 but occurring as early as after the first cycle or second cycle. In one study, of the 75% of patients who had developed grade 2 nail changes, 68% had received more than 4 cycles of treatment. Concomitant, rather than sequential treatment with docetaxel was associated with more nail changes.

Most of the nail changes that have occurred in studies have tended to be grade 1-2, but in a few studies as much as grade 3 or grade 4. Certain combinations of chemotherapy drugs are also associated with more severe nail destruction than others such as docetaxel and transtuzumab and dose-dense docetaxel followed by dose dense doxorubicin / cyclophosphamide. Not surprisingly, nail toxicity may impact on a patient's quality of life, particularly in females and may affect body image, pain, and function, any or all of which has a wider impact on the individual's normal daily activities. In one study, more than two-thirds of the sample who developed changes (86.8%) were significantly limited in activities of daily living. A retrospective study of 425 medical notes, based in the SERIES clinic in New York, examined the range of dermatological toxicities on quality of life (QoL) using the Skindex-16. This tool measured 3 separate domains: symptoms, emotional and function. The authors found 9.2% incidence of nail toxicities, with 32 cases where the individual possessed 3 or more different or associated dermatological toxicities. These identified patients had significantly higher symptom, emotional and function scores than those who had less than three toxicities.

There are reports that nail changes resolve over time, usually after discontinuation or completion of treatment. However, there were a few reports where only partial resolution occurred and residual nail problems persisted. There remains poor understanding of the pathogenesis of nail damage.

It has been demonstrated all 20 participants in a study of patients with metastatic breast cancer had only partial response, irrespective of severity or type of nail change (50% grade 1 and 25% grade 2). One study described a case study of a 66 year old male who developed a grade one, taxane-induced nail problem as persisting for months after completion of treatment but which did eventually improve over time. A further case report of a female who developed hyperpigmentation and sub-ungual haemorrhage after 2 of 4 cycles of docetaxel had residual problems after 12 months of discontinuation of treatment, developing a fungal paronychia which necessitated removal of the nail. An earlier case study demonstrated the gradual resolution of nail conditions despite continuation of treatment. The findings thus far indicate that early recognition is imperative to alleviate symptoms and complete treatment.

The use of filgastrim and/ or erythropoietin prophylactically, prior to treatment, appears to reduce not only the rate of febrile neutropenia but also reduces nail changes and increases compliance with treatment and improvement in quality of life.

In the studies reviewed, prior to trial intervention usual advice to patients receiving taxane therapy is to use a nail hardener at the first sign of nail weakness, keep nails dirt-free, use nail polish, avoid oil baths and wear gloves during household tasks which involve soaking the hands in water. Others suggest that nail changes in individuals receiving taxanes and anthracyclines may be precipitated by sunlight or UV exposure. It has been reported that one patient on weekly paclitaxel for intra-ductal breast cancer who developed both photo-distributed erythema and onycholysis after sun exposure to the affected area and reports associated photosensitivity conditions in nine female oncology patients in total. Therefore, there is some evidence that the use of a nail covering, or UV protective, may at least provide some protection.

Patients have searched for products that may help prevent deterioration of their nails while on chemotherapy treatment. OnicoLife drops are available to purchase online and anecdotally, patients receiving chemotherapy have reported this product reduced soreness, ridging and detachment from the nail bed. The active ingredient in this product is Adelmidrol, a semisynthetic derivative of azelaic acid and analogue of the anti-inflammatory compound palmitoylethanolamide (PEA), which has shown efficacy in the local topical treatment of pain and inflammation. However there is no current evidence based research to support the use with breast cancer patients receiving taxane based chemotherapy.

Vascular abnormalities that predispose to nail changes have also been considered as a way to manage occurrence using cooling interventions. One study used a frozen glove to reduce nail problems, which was then extended to the use of frozen socks in a further study, with significant benefits in both studies. Both studies used the right hand/ foot for the intervention and the left hand or foot as the control. However, no information was provided as to the site of venous access in relation to the intervention and/or if avoidance of the dominant hand was ever considered. The only caveat to using a frozen glove during treatment is therefore venous access problems, and some patients were not able to wear the glove for a predetermined period due to cold intolerance.

Rationale:

Nail problems pose substantial problems for patients with breast cancer undergoing chemotherapy in terms of quality of life. It is a difficult challenge for health care professionals to manage and provide advice, mainly due to the lack of evidence on effective solutions. There is a need to look at the options that may have potential benefit to patients, including toxic-free formulation of dark nail polish and OnicoLife drops ® which appear to be useful, however, there is no research based evidence to support their use.

ELIGIBILITY:
Inclusion Criteria:

* women over the age of 18 years who have been diagnosed with a breast cancer.
* must be receiving adjuvant or neo-adjuvant Taxotere chemotherapy for breast cancer.
* participants must be fluent English speakers to be eligible to take part, as there are no resources or additional funding for translators or interpreting services.
* Participants must provide informed consent.

Exclusion Criteria:

* Male patients with a diagnosis of breast cancer
* Patients who are non-fluent English speakers
* Patients with a known hypersensitivity reaction to nail/ relevant cosmetic products
* Previous treatment with taxane chemotherapy with the last two years
* Patients with only one upper limb.
* Patients with a neurological deficit to the upper limb (eg, stroke affecting one side)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Nail Assessment Scale | 6 months
  Evaluate nail interventions (nail polish + standard care Vs Onicolife drops + standard care Vs Standard Care only) that may prevent or minimise the occurrence and severity of nail problems measured using the NToX-G12 (Nail Assessment Scale).
Adverse Events | 6 months
  Evaluate nail interventions (nail polish + standard care Vs Onicolife drops + standard care Vs Standard Care only) that may prevent or minimise the occurrence and severity of nail problems measured using Common Terminology Criteria for Adverse Events v3.0 (CTC-AE v3).

SECONDARY OUTCOMES:
Quality of Life - NToX-QoL Health related quality of life questionnaire | 6 months
  Evaluate any change in the patient's quality of life, in relation to nail problems occurring, as measured using the NToX-QoL (quality of life questionnaire).
Quality of Life - EQ-5D-5L Health related quality of life questionnaire | 6 months
  Evaluate any change in the patient's quality of life, in relation to nail problems occurring, as measured using the EQ-5D-5L (quality of life questionnaire)
Quality of Life-nail grade severity relationship | 6 months
  Assess collected data for any correlating relationship between nail grade severity (measured using NToX-G12 - outcome measure 1) and qualify of life (measured using NToX-QoL - outcome measure 3).

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Morrison, Phd, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Beatson Oncology Centre, Glasgow, United Kingdom